CLINICAL TRIAL: NCT03933371
Title: Risk Factors of Inadequate Bowel Cleansing in Colon Capsule Endoscopy
Brief Title: Predictors of Poor Bowel Cleansing and Capsule Endoscopy (CEPREDICT)
Acronym: CEPREDICT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitario de Canarias (Other)
Responsible Party: Sponsor
Other Study IDs: CEPREDICT
Record Dates: First submitted 2019-04-28; First posted 2019-05-01 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Colon Adenoma
Keywords: colonoscopy; capsule; Cleansing
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Colon Capsule Endoscopy — The capsule endoscopy will be ingested by the participant. This device captures images along the large bowel. This images are stored in an external memory and afterwards they are downloaded in a computer

SUMMARY:
The main purpose of the study is to determine risk factors of poor bowel cleansing in patients referred for colon capsule endoscopy (CCE) examination. Patients will be prepared with polyethylene glycol (PEG), and a booster by using oral low volume sodium phosphate (NaP) and sodium-amidotrizoate and meglumine-amidotrizoate (Gastrografin ®) The investigators also will try to design a predictive score of poor bowel cleansing and to validate the Bowel cleansing score designed by Leighton and modified by Spada

DETAILED DESCRIPTION:
As in conventional colonoscopy, colon cleansing is essential to achieve a quality examination through the colon capsule endoscopy. The CCE also presents additional difficulties due to the inability to distend the walls of the colon, aspirate liquid and debris and wash. These reasons make that the colonic preparation should be even more effective when the exploration is going to be performed by CCE than with the conventional colonoscopy. Using a combination of PEG, sodium phosphate and bysacodil suppository achieves at least 80% of well-prepared CCE. The rate of CCE with inadequate preparation according to different studies ranges from 12% to 34% . It has recently been suggested that the addition of a water-soluble contrast agent such as Gastrografin® commonly used in different radiological tests could improve cleaning.

Although, predictive factors of poor bowel cleansing in outpatient conventional colonoscopy are well-known, currently, there are no studies that evaluate the independent predictive factors of poor colonic preparation in patients who undergo a CCE. The investigation of the predictive factors of poor colonic preparation in these patients, following the current recommendations can be of great interest to identify those patients with greater difficulties in obtaining an acceptable cleaning quality.

The researchers will offer to participate in the study to patients scheduled for CCE who meet all the inclusion criteria and none of the exclusion criteria. The researchers will explain the purpose of the study and will ask to sign the informed consent. They will give verbal and written information on the diet and the bowel cleansing solution to be taken. The bowel cleansing quality following Spada Bowel Preparation Scale will be assessed by the endoscopist The aim of this study is to figure out the risk factors of bowel cleansing of inadequate bowel preparation in patients referred for colon capsule endoscopy.

A maximum of 8 variables in the multivariate analysis will be included. Considering a percentage of poor preparation of 20%, the inclusion of 350 patients will be necessary. A maximum of 15% of losses will be considered, so the final sample size will be 403 patients.

A univariate and multivariate analysis will be carried out to determine those factors associated with a lack of progression from capsule to rectum and accelerated progression. For the first of these objectives, well prepared colonoscopies but in which the rectum was not identified (identification of the hemorrhoidal plexus) will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients referred for colon capsule endoscopy

Exclusion Criteria:

* Ileus, intestinal obstruction, megacolon.
* Poorly controlled hypertension (HTAS> 180 HTAD> 100).
* Terminal renal failure (pre-dialysis or dialysis).
* Congestive heart failure (NYHA III-IV).
* Acute liver failure.
* Severe psychiatric illness.
* Dementia with difficulty in the intake of the preparation.
* Pregnancy or breastfeeding.
* Refusal to participate in the study.
* Inability to follow the instructions.
* Alergies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred for colon capsule endoscopy meeting inclusion and exclusion criteria will be included in the study. Spanish hospitals with the availability of colon capsule endoscopy will be invited to participate in the study
Sampling Method: Probability Sample
Enrollment: 403 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Colon cleansing | [Time frame: 20 months][Designated as safety issue: No]
  Quality of bowel cleansing assessed by the Spada Bowel Preparation Scale. Cleansing is classified from 1 ( no preparation) to 4 (excellent preparation) in each of the 4 segments of the colon (proximal colon, transverse colon, distal colon and rectum)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Z Gimeno Garcia, MD, PhD, Principal Investigator — Hospital Universitario de Canarias

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Spada C, Hassan C, Munoz-Navas M, Neuhaus H, Deviere J, Fockens P, Coron E, Gay G, Toth E, Riccioni ME, Carretero C, Charton JP, Van Gossum A, Wientjes CA, Sacher-Huvelin S, Delvaux M, Nemeth A, Petruzziello L, de Frias CP, Mayershofer R, Amininejad L, Dekker E, Galmiche JP, Frederic M, Johansson GW, Cesaro P, Costamagna G. Second-generation colon capsule endoscopy compared with colonoscopy. Gastrointest Endosc. 2011 Sep;74(3):581-589.e1. doi: 10.1016/j.gie.2011.03.1125. Epub 2011 May 20. PMID 21601200
- [Result] Alarcon-Fernandez O, Ramos L, Adrian-de-Ganzo Z, Gimeno-Garcia AZ, Nicolas-Perez D, Jimenez A, Quintero E. Effects of colon capsule endoscopy on medical decision making in patients with incomplete colonoscopies. Clin Gastroenterol Hepatol. 2013 May;11(5):534-40.e1. doi: 10.1016/j.cgh.2012.10.016. Epub 2012 Oct 16. PMID 23078891
- [Result] Spada C, Hassan C, Galmiche JP, Neuhaus H, Dumonceau JM, Adler S, Epstein O, Gay G, Pennazio M, Rex DK, Benamouzig R, de Franchis R, Delvaux M, Deviere J, Eliakim R, Fraser C, Hagenmuller F, Herrerias JM, Keuchel M, Macrae F, Munoz-Navas M, Ponchon T, Quintero E, Riccioni ME, Rondonotti E, Marmo R, Sung JJ, Tajiri H, Toth E, Triantafyllou K, Van Gossum A, Costamagna G; European Society of Gastrointestinal Endoscopy. Colon capsule endoscopy: European Society of Gastrointestinal Endoscopy (ESGE) Guideline. Endoscopy. 2012 May;44(5):527-36. doi: 10.1055/s-0031-1291717. Epub 2012 Mar 2. PMID 22389230
- [Result] Spada C, Hassan C, Costamagna G. Colon capsule endoscopy. Gastrointest Endosc Clin N Am. 2015 Apr;25(2):387-401. doi: 10.1016/j.giec.2014.11.007. Epub 2015 Jan 28. PMID 25839692